CLINICAL TRIAL: NCT06394869
Title: Cystoscopic REDuction In BLadder Evaluations for Microhematuria - A Prospective Randomized, Controlled, Clinical Utility Study for Evaluation of Microhematuria (The CREDIBLE Study)
Brief Title: Study to Assess the Impact of the Urine Test Cxbladder Triage Plus on the Number of Cystoscopies Performed on Patients With Invisible Blood in Their Urine.
Acronym: CREDIBLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Edge Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CXB/2024/CREDIBLE
Record Dates: First submitted 2024-04-21; First posted 2024-05-01 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hematuria - Cause Not Known
Keywords: microscopic hematuria; microhematuria; urothelial carcinoma; bladder cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Arm (Experimental): The site will receive the Cxbladder Detect+ result and the urologist study investigator discuss it with the patient before making a shared decision whether or not to proceed with cystoscopy.
  Interventions: Diagnostic Test: Cxbladder Triage Plus
- Control arm (No Intervention): Neither the site nor the patient will receive the Cxbladder Detect+ result. The decision whether or not to proceed with cystoscopy will be made following standard of care.

INTERVENTIONS:
Diagnostic Test: Cxbladder Triage Plus — Cxbladder Triage Plus is a lab developed, test that is using RNA and DNA biomarkers in the urine to assess the likelihood of the presence of urothelial carcinoma in the bladder.
  Arms: Test Arm

SUMMARY:
This study includes adult patients who see a urologist because of blood in their urine. The amount is so small it can only be seen with a microscope. This is called microhematuria. There can be many reasons for microhematuria. One of them is bladder cancer. While bladder cancer is one of the biggest worries, it is only found in few of these patients.

Most microhematuria patients will have a cystoscopy to look inside the bladder. During a cystoscopy, a small camera is inserted into the bladder. This is done through the urethra, the tube that passes urine from the bladder to the outside. In some patients it can cause pain or anxiety. Not all patients have a cystoscopy. Those that don't, usually return for a urine sample within 6 months. This is done to check if there is still blood in their urine.

This study is conducted to find out if the use of "Cxbladder Triage Plus" changes the number of cystoscopies in microhematuria patients. Cxbladder Triage Plus is also called "Triage Plus". It is a lab test that was developed to check how likely urothelial carcinoma is present in the bladder. Urothelial carcinoma is by far the most common type of bladder cancer. For the test, the patient voids some urine into a cup. A laboratory then checks the urine of specific genetic material. Abnormalities can be a sign of urothelial carcinoma. The result indicates if the urine is more like most normal urine or more like that of urothelial carcinoma patients.

The study is done to find out how Triage Plus changes the number of cystoscopies. Study participants first void urine into a cup. The urine is used for the Triage Plus test. The patients are then assigned to one of two groups. The assignment is random. This means the nobody can influence the assignment. The chance to be assigned to either group is the same. In the test group, the urologist will receive the Triage Plus result and discuss it with the patient. Together they decide whether to do a cystoscopy. In the control group, the urologist will not receive the Triage Plus result. The patient will also not get the result. The urologist and patient will follow standard of care to decide whether to do a cystoscopy.

For test group patients, the study gives a recommendation whether to proceed with cystoscopy. It is based on the patient's Triage Plus result. The urologist and patient do not need to follow the recommendation. If the urologist does not follow it, they will complete a survey. The survey has only one question. It is asking for the reasons of the decision.

After making their decision, patients will follow the chosen pathway. Data on the performed procedures are collected. The diagnosis will also be documented. Data will be collected for up to about 9 months.

To see how Triage Plus changes the number of cystoscopies, these will be counted in each group and then compared.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is referred for assessment of microhematuria (MH) with presentation confirmed by urine microscopy of 3 or more red blood cells per high powered field (RBC/HPF) (documented by the referring physician or at the investigator site) within 6-months of enrollment.
2. Physically able to provide a voided urine sample from a bladder that has not been surgically altered.
3. Able to give informed, written consent.
4. Able and willing to comply with study requirements.
5. Must be 19 or the legal age of consent in the jurisdiction in which the study is taking place to 88 years of age inclusive, at the time of signing the informed consent.
6. Ability to comprehend written and spoken English sufficiently to independently follow all study procedures. Or ability to comprehend Spanish with access to an English-Spanish interpreter for all study related verbal instructions and discussions.

Exclusion Criteria:

1. Prior history of bladder malignancy.
2. Prior history of upper tract UC or prostatic urethral UC.
3. Gross hematuria within the last twelve months (reported in patient's records and/or during patient's interview)
4. Reconstructed or diverted bladder (e.g., bladder augmentation, ileal conduit, Indiana pouch)
5. Indication to recommend cystoscopy other than MH (e.g., bothersome benign prostatic hyperplasia symptoms and desires a procedure, weak stream with concerns for urethral stricture).
6. Cystoscopy contraindicated due to another condition or anatomy.
7. History of pelvic radiation.
8. Currently receiving systemic chemotherapy or has had systemic chemotherapy within the last 6 weeks.
9. History of schistosomiasis.
10. History of chronic (>3 months) indwelling Foley catheter or chronic (>3 months) bladder stones.
11. Known current pregnancy

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Cystoscopy rate | 3 months from the decision to perform or not perform cystoscopy.
  Difference in the proportion of cystoscopies performed in each arm.

SECONDARY OUTCOMES:
Rate of imaging procedures | 3 months from the decision to perform or not perform cystoscopy.
  Sub-analyses on AUA risk categories for primary and secondary objectives

OTHER OUTCOMES:
Detection of urothelial carcinoma (UC) | At the end of the current investigation, i.e. when a diagnosis was made or it was decided not to perform diagnostic procedures other than surveillance. Expected within approximately 120 days after sampling.
  Difference in the proportion of UCs found in each arm.
Cxbladder Triage Plus performance and test negative rate. | At the end of the current investigation, i.e. when a diagnosis was made.
  Number of false positive, true positive, false negative and true negative test results when comparing the Triage Plus result to the results of histopathologically confirmed cystoscopy.
Persistent hematuria. | At urinalysis 90-180 days (of the decision to proceed with surveillance)
  Rate of persistent hematuria in patients choosing surveillance.
Physician rationale | After reviewing the Detect+ result and giving their recommendation, before cystoscopy (if applicable). Expected once and within 90 days of sampling
  Physician-reported reasons for not following the study recommended pathway based on the Detect+ result.
Patient rationale | After discussing the Detect+ result with the investigator, before cystoscopy (if applicable). Expected once and within 90 days of sampling .
  Patient-reported reasons for not following the investigator recommended pathway.
Imaging Rates | 3-months prior to 6-months post enrollment
  Change in imaging rates between arms

CONTACTS AND LOCATIONS:
Overall Officials: Tony Lough, PhD, Study Chair — Pacific Edge Limited
Locations (15):
- United States (15):
  - Urology Centers of Alabama, Homewood, Alabama
  - Urology Associates of Mobile, Mobile, Alabama
  - Advanced Urology Institute - Daytona Beach, Daytona Beach, Florida
  - Urologic Specialists of Northwest Indiana, Merrillville, Indiana
  - Southern Urology, Lafayette, Louisiana
  - Chesapeake Urology Research Associates, Hanover, Maryland
  - Summit Health, Voorhees Township, New Jersey
  - Albany MED Health System, Albany, New York
  - Integrated Medical Professionals, New York, New York
  - Premier Medical Group of the Hudson Valley, P. C., Poughkeepsie, New York
  - Penn State Medical Center, Urology Research, Hershey, Pennsylvania
  - Urology Associates, P. C., Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No